CLINICAL TRIAL: NCT06371235
Title: Study of the Transmission of Anti-interferon Type 1 Alpha Autoantibodies From Mother to Child Via the Placental Barrier
Acronym: Pregiferon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CerbaXpert (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A00739-38
Record Dates: First submitted 2024-04-04; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Woman Suffering From a Pathology Frequently Associated With the Presence of These Anti-autoantibodies Type-I Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnant women (Other): Pregnant woman over 18 years old
  - Woman whose gestational age is less than 30 weeks
  Interventions: Other: Pregiferon

INTERVENTIONS:
Other: Pregiferon — This Study aims to study the transmission of anti-interferon alpha autoantibodies from mother to child viaplacental barrier

SUMMARY:
The main objective of the study is to evaluate the frequency of placental transfer of self-Ab directed against the mother's IFN alpha in the newborn, in all women suffering from a pathology frequently associated with the presence of these autoantibodies and in those seropositive during the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman over 18 years old
* Woman whose gestational age is less than 30 weeks.
* Having agreed to carry out an assay of anti-IFN alpha IgG auto-Ac before 30 weeks
* Give birth in the inclusion center
* Suffering from a pathology frequently associated with the presence of these anti-autoantibodies IFN alpha (lupus, severe COVID-19, myasthenia gravis, incontinentia pigmenti, hypoparathyroidism, adrenal insufficiency, diffuse candidiasis, Biermer's disease, dysthyroidism, type 1 diabetes, celiac disease, auto-thyroid disease immune system such as Graves' disease, Hashimoto's thyroiditis) or knowing its positive anti-IFN alpha autoantibody status
* Affiliated with the Social Security system

Exclusion Criteria:

* Patient who underwent a blood transfusion less than 2 months ago
* Patient who received an organ transplant
* Patient undergoing immunotherapy, stem cell therapy and/or other malignancy maternal, under heavy treatment (chemotherapy) less than 6 months before inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of placental transfer of self-Ab directed against IFN alpha from mother to newborn. | 30 months
  A placental transfer will be defined by the presence of anti-IFN alpha IgG auto Ab in the blood.
  of the umbilical cord. The transfer frequency will be calculated with its overall 95% confidence interval and by pathology (lupus, severe COVID-19, myasthenia gravis, incontinentia pigmenti, hypoparathyroidism, adrenal insufficiency, diffuse candidiasis, Biermer's disease, dysthyroidism, type 1 diabetes, celiac disease, autoimmune thyroid disease such such as Graves' disease, Hashimoto's thyroiditis), in HIV-positive women by pathology (lupus, severe COVID-19, myasthenia gravis, incontinentia pigmenti, hypoparathyroidism, adrenal insufficiency, diffuse candidiasis, Biermer's disease, dysthyroidism, type 1 diabetes, celiac disease, autoimmune thyroid disease such as Graves' disease, Hashimoto's thyroiditis), in HIV-positive women.